CLINICAL TRIAL: NCT04283370
Title: A Study Protocol Randomised Feasibility Trial Comparing a Home Rehabilitation Program Versus e-Health Program on Disability, Pain, Fear of Movement, Quality of Life and Spinal Mobility in Non-specific Low Back Pain
Brief Title: A Study Protocol Comparing a Home Rehabilitation Program Versus e-Health Program in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC-0185-2017
Record Dates: First submitted 2020-02-10; First posted 2020-02-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Low-back Pain
Keywords: low back pain; electroanalgesia; exercise program; e-health; Randomized Controlled Trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home rehabilitation program (Experimental): It consists in a home rehabilitation program. Patients will recieve electroanalgesia with TENS and an exercise program following the McKenzie method. At first and second sessions, patients will be instructed on how to use electroanalgesia and how to perform the exercises. Then, patients will perform the therapy at home. Patients will perform the treatment 3 times per week, for 4 weeks, with a total of 24 sessions
  Interventions: Other: Home Rehabilitation Program
- e-Health program (Active Comparator): It consists in a support system for the treatment of chronic low back pain based on web technologies. The system can register a subject and provide a treatment of electroanalgesia and exercise through the Mckenzie method. Video applications of electroanalgesia and exercises will be shown to patients who use their computer or mobile device to access the platform through the Internet. The treatments will be recommended by the system based on the database that is configured to accommodate the application of electroanalgesia and McKenzie exercises based on the diagnosis according to the McKenzie method.patients will perform the treatment 3 times per week, for 4 weeks, with a total of 24 sessions
  Interventions: Other: e-Health program

INTERVENTIONS:
Other: Home Rehabilitation Program — It consists in a home rehabilitation program performing electroanalgesia and an exercise program following the Mckenzie method. Patients will be instructed in the use of the TENS device using 5x9cm electrodes at the bilateral paravertebral level, the patients that present radicular pain, the electrodes will be placed in the path of the affected nerve. The realization of exercises will be through the application of an Mckezie protocol. The duration will be the same as that used to carry out the Mckenzie protocol. Mckenzie exercises are designed to make changes in the internal components periarticular of the spine.
  Arms: Home rehabilitation program
Other: e-Health program — It consists in an e-Health rehabilitation program through a web platform performing electroanalgesia and an exercise program following the Mckenzie method. Patients will be instructed in the use of the TENS device using 5x9cm electrodes at the bilateral paravertebral level, the patients that present radicular pain, the electrodes will be placed in the path of the affected nerve. The realization of exercises will be through the application of an Mckezie protocol. The duration will be the same as that used to carry out the Mckenzie protocol. Mckenzie exercises are designed to make changes in the internal components periarticular of the spine.
  Arms: e-Health program

SUMMARY:
The aim of this randomized controlled trial is to evaluate the feasibility and effectiveness of providing an e-Health rehabilitation program through a web platform performing electroanalgesia and an exercise program following the McKenzie Method for patients with chronic low back pain in primary care, compared with the same home rehabilitation program but without the support of an electronic program.

DETAILED DESCRIPTION:
A double blind clinical trial will be developed in a sample of 80 subjects with chronic low back pain. Patients will receive 3 weekly sessions of electroanalgesia and an exercise program for 8 weeks, for a total of 24 sessions. The aim is to analyze the effectiveness of a home rehabilitation program vs a web platform program on disability, pain, fear of movement, quality of life, resistance of the trunk flexors, lumbar mobility in flexion and muscular electrical activity.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ≥ 3 months.
* Age between 30 and 67 years old.
* Score ≥ 4 points on the Roland Morris Disability Questionnaire.
* Not being receiving physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis.
* Diagnosis of spondylolisthesis.
* Diagnosis of fibromyalgia.
* Treatment with corticosteroids or oral medication in recent weeks.
* History of spine surgery.
* Contraindication of analgesic electrical therapy.
* Have previously received a treatment of electrical analgesia or exercise.
* Central or peripheral nervous system disease.
* Agoraphobia

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline the acceptability and demand of the e-Health intervention for patients and physiotherapists in comparison with the home rehabilitation program for the optimization of their design, development and delivery | At baseline, immediate post-treatment and 6 months
  The extent to which participants who have received the intervention through a web application consider that the content and support materials (web application and initial learning sessions) are appropriate and satisfactory to obtain the expected results.The extent to which the physiotherapists who have administered the intervention consider that the training, content and support materials are appropriate.Brief questionnaire developed for this trial* 10-items Patients rate their acceptability and demand of treatment received and trial participation, including the burden of outcome measure completion. Measured with 10-point numeric rating scales ranging from not at all satisfactory to extremely satisfactory
Change from baseline the feasibility of the trial procedures | At baseline, immediate post-treatment and 6 months
  The extent to which participants believe that their eligibility, outcome measures, follow-up and intervention by the physiotherapist have been satisfactory.
  The extent to which physiotherapists who have participated in the trial consider recruitment, outcome measures, evaluation follow-ups and appropriate and satisfactory intervention procedures.Brief questionnaire developed for this trial* 4-items Measured with 10-point numeric rating scales ranging from not at all helpful to extremely helpful
Change from baseline adaptation of the e-Health intervention and the trial procedures for to randomized clinical trial definitive | At baseline, immediate post-treatment and 6 months
  The extent to which the content of the e-health intervention, support materials and learning classes should be modified to improve their acceptability and implementation for a future definitive trial The extent to which recruitment, follow-up procedures and the number and outcome measures should be modified during / at the end of the trial to improve its acceptability and implementation for a definitive future trial.Brief questionnaire developed for this trial* 11-items Measured using yes/no responses

SECONDARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire | At baseline, at 8 weeks and at 6 months
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.Ranging from 0 points- better to 24 points- worse disability
Change from baseline in disability. Oswestry Low Back Pain Disability Idex. | At baseline, at 8 weeks and at 6 months
  It has 10 items associated to activities of daily living, each ítem has a puntuation fron 0 to 5 points.The higher scores mean a worse outcome
Change from baseline in pain intensity. Visual analogue scale. | At baseline, at 8 weeks and at 6 months
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain.Range from no pain 0 to maximum pain 10 points
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline, at 8 weeks and at 6 months
  Is a 17-item questionnaire that measures the fear of movement and (re)injury.Patient rate beliefs about their kinesiophobia on a 4-point scale ranging from strongly disagree to strongly agree.
Change from baseline on Quality of Life. SF-36 Health questionnaire. | At baseline, at 8 weeks and at 6 months
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.The higher the score, the higher the quality of life
Change from Mcquade Test. | At baseline, at 8 weeks and at 6 months
  It measures the isometric endurance of trunk flexion muscles in seconds.
Change from baseline in lumbar mobility flexion. | At baseline, at 8 weeks and at 6 months
  For the quantification of lumbar flexion an angular inclinometer is used (Fleximeter UM 8320-3 RJ Code Research Institute, Brazil).
Changes from baseline in Lumbar electromyography. | At baseline, at 8 weeks and at 6 months
  The degree of electromyographic activation of the lumbar paravertebral musculature will be carried out by using a set of electrodes of 3x7 dimensions that will be applied uniformly in the lumbar region from the spinal level from L2 to L5.
Change from baselina in range of motion and lumbar segmental mobility | At baseline, at 8 weeks and at 6 months
  This variable is quantified using the SpinalMouse ® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagittal spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro-Sánchez, PhD, Principal Investigator — Almeria University
Locations (1):
- Almeria University, Almería, Spain

REFERENCES:
- [Background] Von Korff M, Moore JC. Stepped care for back pain: activating approaches for primary care. Ann Intern Med. 2001 May 1;134(9 Pt 2):911-7. doi: 10.7326/0003-4819-134-9_part_2-200105011-00016. PMID 11346328
- [Background] Schaafsma FG, Whelan K, van der Beek AJ, van der Es-Lambeek LC, Ojajarvi A, Verbeek JH. Physical conditioning as part of a return to work strategy to reduce sickness absence for workers with back pain. Cochrane Database Syst Rev. 2013 Aug 30;2013(8):CD001822. doi: 10.1002/14651858.CD001822.pub3. PMID 23990391
- [Background] Becker A, Held H, Redaelli M, Strauch K, Chenot JF, Leonhardt C, Keller S, Baum E, Pfingsten M, Hildebrandt J, Basler HD, Kochen MM, Donner-Banzhoff N. Low back pain in primary care: costs of care and prediction of future health care utilization. Spine (Phila Pa 1976). 2010 Aug 15;35(18):1714-20. doi: 10.1097/brs.0b013e3181cd656f. PMID 21374895
- [Background] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758
- [Background] Elfering A, Semmer N, Birkhofer D, Zanetti M, Hodler J, Boos N. Risk factors for lumbar disc degeneration: a 5-year prospective MRI study in asymptomatic individuals. Spine (Phila Pa 1976). 2002 Jan 15;27(2):125-34. doi: 10.1097/00007632-200201150-00002. PMID 11805656
- [Background] Haladay DE, Miller SJ, Challis J, Denegar CR. Quality of systematic reviews on specific spinal stabilization exercise for chronic low back pain. J Orthop Sports Phys Ther. 2013 Apr;43(4):242-50. doi: 10.2519/jospt.2013.4346. Epub 2013 Jan 14. PMID 23321935
- [Background] Palacin-Marin F, Esteban-Moreno B, Olea N, Herrera-Viedma E, Arroyo-Morales M. Agreement between telerehabilitation and face-to-face clinical outcome assessments for low back pain in primary care. Spine (Phila Pa 1976). 2013 May 15;38(11):947-52. doi: 10.1097/BRS.0b013e318281a36c. PMID 23238489
- [Background] Descarreaux M, Normand MC, Laurencelle L, Dugas C. Evaluation of a specific home exercise program for low back pain. J Manipulative Physiol Ther. 2002 Oct;25(8):497-503. doi: 10.1067/mmt.2002.127078. PMID 12381971
- [Background] Petersen T, Kryger P, Ekdahl C, Olsen S, Jacobsen S. The effect of McKenzie therapy as compared with that of intensive strengthening training for the treatment of patients with subacute or chronic low back pain: A randomized controlled trial. Spine (Phila Pa 1976). 2002 Aug 15;27(16):1702-9. doi: 10.1097/00007632-200208150-00004. PMID 12195058
- [Background] Khadilkar A, Odebiyi DO, Brosseau L, Wells GA. Transcutaneous electrical nerve stimulation (TENS) versus placebo for chronic low-back pain. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003008. doi: 10.1002/14651858.CD003008.pub3. PMID 18843638